CLINICAL TRIAL: NCT01535352
Title: Depressed Mothers in Rural Areas: Web-Facilitated Cognitive Behavioral Treatment
Acronym: Mom-NetRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH091199-02 (NIH)
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Maternal Care Patterns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Internet-facilitated CBT (Experimental): Participants in the randomized trial will be 300 mothers of 3-5 year old children recruited through Head Start (HS) classrooms and screened for the presence of major or minor depression. Subsequent to the pre-intervention assessment, participants will be randomized, with an allocation ratio of 1:1, to either the Mom-Net (MN) intervention or facilitated usual care (FUC) condition. Participants in the MN condition will receive the Mom-Net intervention. The Mom-Net program is an internet-facilitated cognitive-behavioral intervention for depression, adapted from the CWDC, and tailored to mothers of young children. Participants in both conditions will receive Booster calls during the follow-up period.
  Interventions: Behavioral: Mom-Net
- Coach-facilitated Treatment as Usual (Active Comparator): Participants in the FUC condition will receive assistance in accessing mental health interventions through community providers that serve low-income individuals. In order to control for the supportive attention provided to mothers in the MN condition by the weekly coach calls, mothers in the FUC condition will receive weekly check-in calls from research staff during the intervention period. Participants in both conditions will receive Booster calls during the follow-up period.
  Interventions: Behavioral: Coach-facilitated Treatment as Usual

INTERVENTIONS:
Behavioral: Mom-Net — The Mom-Net intervention is an internet-facilitated cognitive-behavioral intervention for depression, adapted from the CWDC, and tailored to mothers of young children. Mom-Net has several core components: 1. A guided course for self-regulated learning of CBT skills. 2. A system of professional support in which coaches provide weekly 15-20 min phone check-ins (coach calls) in order to encourage and facilitate progress through the intervention and respond rapidly to participant queries and emergencies. In this regard, coaches benefited from: a) a 'behind the scenes" administration page on the website that enabled them to track participants' progress through the intervention and use this information to tailor coaching sessions; and b) an automated system for alerting coaches/supervisors when participants were in crisis. 3. A coach-moderated bulletin board that approximated the social support provided by group administration.
  Arms: Internet-facilitated CBT
Behavioral: Coach-facilitated Treatment as Usual — Participants in the facilitated usual care (FUC) condition will receive assistance in accessing mental health interventions through community providers that serve low-income individuals. In order to control for the supportive attention provided to mothers in the MN condition by the weekly coach calls, mothers in the FUC condition will receive weekly check-in calls from research staff during the intervention period. Participants in both conditions will receive Booster calls during the follow-up period.
  Arms: Coach-facilitated Treatment as Usual

SUMMARY:
Low income mothers of young children represent a disadvantaged group who are at exceptional risk for depressive syndromes and who have increasingly limited access to mental health services. The proposed project is designed to evaluate Mom-Net, an internet-facilitated cognitive-behavioral(CBT) intervention for depression, adapted from Lewinsohn's Coping with Depression Course, and tailored to mothers of young children. Mom-Net, which was developed and piloted in an recently completed NIMH-funded investigation (MH070426), was designed to overcome the substantial barriers to treatment participation that exist for mothers experiencing economic hardship and those in rural communities. Though the pilot trial demonstrated that the program was very effective in reducing depressive symptoms and related difficulties, it was conducted under the 'idealized' conditions typical of initial intervention tests (e.g., computers and internet connections were supplied to all participants; access to the internet was provided by a single browser; coaches who provided weekly phone support were research staff, and initial recruitment and motivational interviews sessions were conducted via home visits to participants). These conditions likely facilitated recruitment and retention of participants, as well as ease and fidelity of treatment delivery. Thus one goal of the current project is to evaluate the intervention under conditions that are closer to those of real-world service providers and recipients. The current project is also intended to provide a more rigorous test of the intervention than did the pilot in a number of ways. Participants in the pilot trial will be 300 mothers of 3-5 year old children recruited through Head Start classrooms and prescreened for the presence of elevated depressive symptoms.Subsequent to the pre-intervention assessment, participants will be randomized to either the intervention or facilitated usual care (FUC) condition. The evaluation of the intervention will focus on maternal depressive symptoms, parenting behavior, and child adjustment. Two follow-up assessments (at 12-month and 24-month intervals) will enable us to examine maintenance of effects. Overall, the investigation will contribute to the evidentiary base regarding the dissemination potential of this empirically-supported intervention, adaptations to which have the potential to enable a greater proportion of the population to access and benefit from it.

DETAILED DESCRIPTION:
The project is designed to evaluate Mom-Net, an internet-facilitated cognitive-behavioral (CBT) intervention for depression, adapted from Lewinsohn's Coping with Depression Course, and tailored to mothers of young children. Mom-Net, which was developed and piloted in a recently completed NIMH-funded investigation (MH070426), was designed to overcome the substantial barriers to treatment participation that exist for mothers experiencing economic hardship and those in rural communities. Though the pilot trial demonstrated that the program was very effective in reducing depressive symptoms and related difficulties, it was conducted under the 'idealized' conditions typical of initial intervention tests (e.g., computers and internet connections were supplied to all participants; access to the internet was provided by a single browser; coaches who provided weekly phone support were research staff, and initial recruitment and motivational interviews sessions were conducted via home visits to participants). These conditions likely facilitated recruitment and retention of participants, as well as ease and fidelity of treatment delivery. Thus one goal of the current project is to evaluate the intervention under conditions that are closer to those of real-world service providers and recipients. The current project is also intended to provide a more rigorous test of the intervention than did the pilot in a number of ways. Participants in this project will be 300 mothers of 3-5 year old children recruited through Head Start classrooms and prescreened for the presence of elevated depressive symptoms. Subsequent to the pre-intervention assessment, participants will be randomized to either the intervention or facilitated usual care (FUC) condition. The evaluation of the intervention will focus on maternal depressive symptoms, parenting behavior, and child adjustment. Two follow-up assessments (at 12-month and 24-month intervals) will enable us to examine maintenance of effects. Overall, the investigation will contribute to the evidentiary base regarding the dissemination potential of this empirically-supported intervention, adaptations to which have the potential to enable a greater proportion of the population to access and benefit from it.

ELIGIBILITY:
Inclusion Criteria:

* Mother of 3-5 year old child(ren)
* Reside in rural community, as defined by RUCA
* Meet DSM IV criteria for major or minor depression based on PHQ-9

Exclusion Criteria:

* Cannot comprehend spoken English
* Being treated for depression at intake

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2012-09; Primary Completion 2016-06 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
PHQ-9 | 4 months, 16 months, 28 months
  Severity of depression

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Options Counseling Services of Oregon, Eugene, Oregon
  - Oregon Research Institute, Eugene, Oregon

REFERENCES:
- [Result] Sheeber LB, Feil EG, Seeley JR, Leve C, Gau JM, Davis B, Sorensen E, Allan S. Mom-net: Evaluation of an internet-facilitated cognitive behavioral intervention for low-income depressed mothers. J Consult Clin Psychol. 2017 Apr;85(4):355-366. doi: 10.1037/ccp0000175. PMID 28333536
- [Result] Seeley JR, Sheeber LB, Feil EG, Leve C, Davis B, Sorensen E, Allan S. Mediation analyses of Internet-facilitated cognitive behavioral intervention for maternal depression. Cogn Behav Ther. 2019 Jul;48(4):337-352. doi: 10.1080/16506073.2018.1513554. Epub 2018 Oct 12. PMID 30311850